CLINICAL TRIAL: NCT06314412
Title: Perineal Rehabilitation: Efficacy of Transcutaneous Posterior Tibial Nerve Stimulation in Patients With Multiple Sclerosis Related Urge Incontinence
Brief Title: Transcutaneous Posterior Tibial Nerve Stimulation in Patients With Multiple Sclerosis Related Urge Incontinence
Acronym: SANS-REHAB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24C211
Record Dates: First submitted 2024-03-04; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Multiple Sclerosis
Keywords: Incontinence; Perineum; Stoller's Afferent Nerve Stimulation; Posterior tibial nerve stimulation
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Multiple Sclerosis (Experimental): Patients with Multiple Sclerosis
  Interventions: Other: Stoller's Afferent Nerve Stimulation (SANS)

INTERVENTIONS:
Other: Stoller's Afferent Nerve Stimulation (SANS) — 15 sessions of SANS (5 sessions/week for 3 weeks)

SUMMARY:
Recently, several studies have investigated the safety and efficacy of the Stoller afferent nerve stimulation (SANS) treatment in Multiple Sclerosis (MS) patients. However, because of the differences among the published protocols (percutaneous versus transcutaneous stimulation, stimulation site, total number of sessions), and the absence of data on the duration of the effect, this treatment is not yet currently included in the rehabilitation programs. The present study aims at evaluating the efficacy of a protocol of SANS in the short- and medium-term follow-up.

The efficacy of the proposed stimulation protocol on the physiological parameters of bladder function will be also investigated.

DETAILED DESCRIPTION:
The primary outcome will be the variation of urinary urgency and incontinence. It will be evaluated by self-reported measuring scales, such as the Overactive Bladder Questionnaire (OAB-q) and the International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) in their Italian forms.

The expected outcome is that the treatment of posterior tibial nerve stimulation will reduce the frequency and the urgency of urination, and urinary incontinence. Moreover, results from the follow-up will allow estimating the duration of the expected outcome.

ELIGIBILITY:
Inclusion Criteria:

* MS diagnosis according to the revised McDonalds criteria. Relapsing-remitting, primary and secondary progressive MS forms are allowed;
* Expanded Disability Status Scale (EDSS) between 2 and 6.5 included;
* MiniMental State Examination ≥ cut off 24/84 by sex/age

Exclusion criteria:

* Any of the following in the month before enrolment: an MS relapse; current corticosteroids therapy because of MS; change in medicines prescribed against fatigue; attending an intensive physical therapy program;
* New or active lesions on a brain or spinal cord MRI scan in the 12 months before the study enrolment;
* Any musculoskeletal disease or any additional neurological disorder
* Urinary infections or surgery in perineal regions
* Skin lesions or carcinoma in situ
* Pregnancy
* Expanded Disability Status Scale (EDSS) ≥ 7;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Measure of variation of incontinence. | Baseline, at 3 weeks after the start of SANS, at 2 months after the end of SANS
  Evaluated by the International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) in the Italian language.
Measure of variation of urinary urgency | Baseline, at 3 weeks after the start of SANS, at 2 months after the end of SANS
  Evaluated by the Overactive Bladder Questionnaire (OAB-q) in the Italian language.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Perucca, MD, Principal Investigator — Istituto Auxologico Italiano
Locations (1):
- Istituto Auxologico Italiano, Milan, Italy